CLINICAL TRIAL: NCT00774527
Title: Randomized Comparison of Cyclophosphamide Versus Cyclophosphamide Plus Fludarabine In Addition To Anti-Thymocyte Globulin for the Conditioning Therapy in Allogeneic Hematopoietic Cell Transplantation for Bone Marrow Failure Syndrome
Brief Title: Comparison of Cy-Atg Vs Cy-Flu-Atg for the Conditioning Therapy in Allo-HCT
Acronym: CyFluCyATG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cooperative Study Group A for Hematology (Network)
Responsible Party: COSAH, Cooperative Study Group A for Hematology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-002
Record Dates: First submitted 2008-10-12; First posted 2008-10-17 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2011-02

CONDITIONS: Bone Marrow Failure Syndromes
MeSH Terms: conditions — Bone Marrow Failure Disorders | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ArmI(CyATG) (No Intervention): •Conditioning therapy will start on day -5 in patients who are randomized to receive Cy+ATG. Hydration with 0.45% NaCl at 6 liters/24 hours will be started on day -5. Cy 50 mg/kg in D5W 200 ml i.v. over 1-2 hours on days -5 to -2 by pump through a central venous catheter
  Interventions: Drug: Cyclophosphamide-fludarabine-anti thymocyte globulin

INTERVENTIONS:
Drug: Cyclophosphamide-fludarabine-anti thymocyte globulin — * Cyclophosphamide 50 mg/kg in D5W 200 ml i.v. over 1-2 hours on days -5 to -2 by pump through a central venous catheter.
  * Fludarabine 30 mg/m2 will be infused intravenously over 30 minutes in D5W 100 ml for 5 consecutive days (days -6 to -2).
  * Thymoglobuline 3 mg/kg in N/S 500-800 mL (less than 0.5 mg/mL) or lymphoglobuline 15 mg/kg in N/S 500-800 mL (less than 2 mg/mL) iv daily at 8 am on days -4 to -2.
  Other Names: CYCLOPHOSPHAMIDE,FLUDARA,ANTI-THYMOCYTE GLOBULINE

SUMMARY:
Randomized comparison of cyclophosphamide versus reduced-dose cyclophosphamide plus fludarabine in addition to anti-thymocyte globulin for the conditioning therapy in allogeneic hematopoietic cell transplantation for bone marrow failure syndrome.

DETAILED DESCRIPTION:
This is a prospective, randomized, non-blind study.

Conditioning therapy will start on day -5 in patients who are randomized to receive Cy+ATG. Hydration with 0.45% NaCl at 6 liters/24 hours will be started on day -5. Cy 50 mg/kg in D5W 200 ml i.v. over 1-2 hours on days -5 to -2 by pump through a central venous catheter. Mesna 12 mg/kg iv push immediately before Cy and 3, 6, 9, and 12 hours after Cy. Thymoglobuline 3 mg/kg in N/S 500-800 mL (less than 0.5 mg/mL) or lymphoglobuline 15 mg/kg in N/S 500-800 mL (less than 2 mg/mL) iv daily at 8 am on days -4 to -2. Premedication for ATG (ALG) will include methylprednisolone 2 mg/kg iv infusion, Tylenol 600 mg po, and Avil 45.5 mg iv push. The doses of cyclophosphamide and ATG (ALG) will be calculated using actual body weight.

Conditioning therapy will start on day -6 in patients who are randomized to receive Cy+fludarabine (FludaraÂ®, Berlex Laboratories, Richmond, CA)+ATG. Fludarabine 30 mg/m2 will be infused intravenously over 30 minutes in D5W 100 ml for 5 consecutive days (days -6 to -2). Thymoglobuline 3 mg/kg in N/S 500-800 mL (less than 0.5 mg/mL) or lymphoglobuline 15 mg/kg in N/S 500-800 mL (less than 2 mg/mL) iv daily at 8 am on days -4 to -2. Premedication for ATG (ALG) will include methylprednisolone 2 mg/kg iv infusion, Tylenol 600 mg po, and Avil 45.5 mg iv push. Hydration with 0.45% NaCl at 6 liters/24 hours will be started on day -3. Cy 50 mg/kg in D5W 200 ml i.v. over 1-2 hours on days -3 to -2 by pump through a central venous catheter. Mesna 12 mg/kg iv push immediately before Cy and 3, 6, 9, and 12 hours after Cy. The doses of cyclophosphamide and ATG (ALG) will be calculated using actual body weight.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bone marrow failure syndrome.
* Written informed consent must be obtained from the patients and donors.
* Patients should have an HLA-identical or one-locus mismatched sibling, family or unrelated donor who is 60 years or less.
* Patients should be 15 years of age or older, but younger than 60 years.
* The performance status of the patients should be 70 or over by Karnofsky performance scale (see Appendix I).
* Patients should not have major illness or organ failure.
* Patients must have adequate hepatic function (bilirubin less than 2 mg/dl, AST and ALT less than three times the upper normal limit).
* Patients must have adequate renal function (creatinine less than 2.0 mg/dl).
* Patients must have adequate cardiac function (ejection fraction > 45% on MUGA scan).
* Patients must not have a psychiatric disorder or mental deficiency severe as to make compliance with the treatment unlikely, and making informed consent impossible.
* Patients must not be in pregnancy.

Exclusion Criteria:

* Patients should have major illness or organ failure

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 82 (Actual)
Dates: Start 2003-03; Primary Completion 2010-02 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of regimen related toxicities | 7 years
  1.1 Compare the regimen related toxicities of two different conditioning regimens, cyclophosphamide (Cy)+anti-thymocyte globulin (ATG) (Cy-ATG) vs. reduced dose of Cy+fludarabine (Flu)+ATG (Cy-Flu-ATG) after allogeneic hematopoietic cell transplantation (allo-HCT).

SECONDARY OUTCOMES:
Secondary end point will be the occurrence of engraftment failure (primary and secondary) | 7years

CONTACTS AND LOCATIONS:
Overall Officials: Kyoo-Hyung Lee, Doctor, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- See also: Cy-ATG vs Cy-Flu-ATG — http://www.google.co.kr